CLINICAL TRIAL: NCT00854646
Title: Phase I Dose Escalation Study of ON 01910.Na With Increasing Duration of an Initial 3-Day Continuous Infusion in Patients With Refractory Leukemia or MDS
Brief Title: Phase I Study of ON 01910.Na in Refractory Leukemia or Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-05
Record Dates: First submitted 2009-02-20; First posted 2009-03-03 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Acute Myelocytic Leukemia; Acute Lymphocytic Leukemia; Chronic Myelocytic Leukemia; Chronic Lymphocytic Leukemia; Myelodysplastic Syndromes
Keywords: ON 01910.Na; refractory; leukemia; myelodysplastic; cell cycle
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes; Leukemia | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ON 01910.Na (Experimental): The starting dose is 650 mg/m2 per day for 3 continuous days every 2 weeks. In successive courses, infusion time may be increased by 1 day up to 7 days every two weeks and/or drug dose may be increased (650, 1050, 1700 mg/m2/day, etc.). After 4 2-week cycles, cycle length may be extended to 3 or 4 weeks. Treatment continues until evidence of disease progression, intolerable adverse events or withdraw of consent.
  Interventions: Drug: ON 01910.Na

INTERVENTIONS:
Drug: ON 01910.Na — The drug is a sterile, concentrated 75mg/mL solution in polyethylene glycol 400, in labeled, sealed glass vials. The Concentrate must be diluted with aqueous infusion solutions (0.9% NaCl, USP and Water for Injection, USP according to instructions) immediately prior to intravenous administration.
  Other Names: Sodium(E)2,4,6trimethoxystyryl-4methoxy-3glycylbenzylsulfone; rigosertib sodium

SUMMARY:
This is an open-label, Phase I study to determine the highest amount of the study drug, ON 01910.Na, that can be safety given to patients with high risk myelodysplastic syndromes (MDS) or refractory leukemias. Patients will receive ON 01910.Na (at a starting dose of 650 mg/m2) intravenously by 3-day continuous infusion once every 2 weeks. Successive courses will use longer infusion times and/or higher doses of the drug until toxicity, effectiveness, or ineffectiveness is recognized. In addition, the amount of drug in the blood will be measured, any antitumor activity will be documented, and the biological effect of ON 01910.Na on cell-cycle pathways will be evaluated in peripheral blood mononuclear cells.

DETAILED DESCRIPTION:
Patients must have histologically documented or cytologically confirmed diagnosis of acute myelocytic leukemia refractory to standard induction treatment, or relapsed after standard therapy; acute lymphocytic leukemia refractory to induction treatment, or relapsed after effective therapy; chronic myelocytic leukemia refractory to imatinib therapy or second line tyrosine kinase inhibition, or relapsed after tyrosine kinase inhibition, in chronic, accelerated, or blastic phase; chronic lymphocytic leukemia refractory to standard therapy, or relapsed in second relapse; a myelodysplastic syndrome (including chronic myelomonocytic leukemia) refractory to azacitidine; and an int-2 or high myelodysplastic syndrome relapsed after a hypomethylating agent. Patients may not be eligible for, or must have declined, bone marrow transplantation or other chemotherapeutic regimens known to produce consistent remissions. Because hematopoietic criteria in leukemia and lymphoma are confounded by the nature of the diseases themselves, there are no hematologic exclusions from treatment. If leukopenia is clinically determined to be attributable to prior treatment, ON 01910.Na treatment may start when the leukocyte count increases on two successive determinations performed at least three days apart. Thrombocytopenia is not a criterion, and patients will be supported with platelet transfusions as clinically necessary. In the absence of leukopenia, a failed prior treatment may be succeeded immediately by entry into study of ON 01910.Na if the leukocyte count is stable or rising, on two successive determinations performed at least three days apart, in the absence of other drug toxicity.

The patient population will involve approximately 12 to 28 patients ≥ 18 years of age in the dose escalation portion of the protocol. All patients must have relapsed or refractory leukemia or poor risk MDS (i.e., int-2 or high risk MDS who have failed standard therapy). They must not be candidates for known regimens or protocol treatments of higher efficacy or priority. Patients with relapsed/refractory leukemia or poor risk MDS must have an ECOG Performance Status of 0, 1, or 2. Patients must have an expected survival, in the opinion of the Investigator, to allow a sufficient observation period for evaluating ON 01910.Na, and meet the eligibility criteria for patients with leukemia or poor risk MDS. After the maximally tolerated dose and the Recommended Phase II Dose (RPTD) and duration are determined, up to 12 additional patients with histologically documented or cytologically confirmed leukemia or poor risk MDS will be added to confirm the appropriateness of the RPTD. Inclusion criteria for the dose confirmation phase will be similar to those of the dose escalation phase of the study, but the ECOG Performance Status must be 0 or 1.

Safety data, including laboratory parameters and adverse events, will be collected for all patients in order to determine the qualitative and quantitative toxicity, and reversibility of toxicity, of ON 01910.Na. Leukemic cells and MDS cells in peripheral blood will be measured on a daily basis during infusion, and at least two times weekly during the following week. If leukemic cells disappear from the blood or blood counts improve as defined by IWG criteria in MDS patients, a bone marrow aspiration will be performed to determine response status in the bone marrow.

All patients may continue therapy for at least six cycles unless rapid disease progression is documented. Patients with an objective clinical response or stable disease can continue up to six more cycles. Further continuation will be determined by the clinical judgment of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically documented or cytologically confirmed diagnosis of acute myelocytic leukemia refractory to standard induction treatment, or relapsed after standard therapy
* Acute lymphocytic leukemia refractory to induction treatment, or relapsed after effective therapy
* Chronic myelocytic leukemia refractory to imatinib therapy or second line tyrosine kinase inhibition, or relapsed after tyrosine kinase inhibition, in chronic, accelerated, or blastic phase
* Chronic lymphocytic leukemia refractory to standard therapy, or relapsed in second relapse
* A myelodysplastic syndrome (including chronic myelomonocytic leukemia) refractory to a hypomethylating agent
* And a int-2 or high myelodysplastic syndrome relapsed after a hypomethylating agent.
* Patients may not be eligible for, or must have declined, bone marrow transplantation or other chemotherapeutic regimens known to produce consistent remissions.
* There are no hematologic exclusions from treatment.
* Patients with prior radiotherapy are eligible unless leukopenia is ascribed to prior radiation treatment, and then entry to study of ON 01910.Na may be initiated when two successive leukocyte counts are rising.
* ECOG Performance Status of 0, 1, or 2 if patient is in the dose escalation phase or 0 or 1 if patient is in the dose escalation phase.
* Patients may have any hematologic parameters without regard to numbers provided that transfusional support is available and the Investigator stipulates that leukopenia is attributable to disease rather than to prior therapy.
* Total bilirubin ≤ 1.5 mg/dL, unless the patient has active hemolysis, or the elevation is secondary to ineffective erythropoiesis.
* Serum creatinine ≤ 1.5 mg/dL, or a calculated creatinine clearance of ≥ 60 mL/min/1.73 m2.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) while in the study. If a woman becomes pregnant or suspects she is pregnant while on study, her treating physician should be informed immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have positive blood cultures until they are afebrile for 3 days on antibiotic therapy which will continue.
* Patients who have leukopenia attributed to prior chemotherapy until two successive leukocyte counts are increasing. Patients with rapidly rising WBC (e.g. >50% increase over the previous day for 3 consecutive days) or WBC > 40 x 109/L.
* Patients who have continuing toxicity other than hematologic from prior therapy until it has resolved to grade 1 or less and will not compromise ON 01910.Na administration.
* Patients who are receiving any other investigational agents or concurrent chemotherapy, radiotherapy, or immunotherapy.
* Patients receiving corticosteroids or colony-stimulating factors may continue on these treatments. These agents will not be introduced if previously not employed.
* Patients with known meningeal infiltration may be included in this clinical trial only if intrathecal therapy and/or radiation has been completed, and cerebrospinal fluid cytology is improved.
* Patients with a history of allergic reactions attributable to compounds of similar chemical or biologic composition to ON 01910.Na.
* Patients should have no major third space fluid accumulation, ascites requiring active medical management including paracentesis, peripheral bilateral edema, or hyponatremia (serum sodium value less than 134 Meq/L).
* Patients with uncontrolled intercurrent illness including, but not limited to uncontrolled ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and nursing women are excluded from this study.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety data, including laboratory parameters and adverse events, will be collected for all patients in order to determine the qualitative and quantitative toxicity, and reversibility of toxicity, of ON 01910.Na. | 2 - 4 months

SECONDARY OUTCOMES:
To investigate the clinical pharmacology of ON 01910.Na including plasma pharmacokinetics, pharmacodynamics and biological effects on cell-cycle pathways. | 2 - 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lewis R. Silverman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Background] Seetharam M, Fan AC, Tran M, Xu L, Renschler JP, Felsher DW, Sridhar K, Wilhelm F, Greenberg PL. Treatment of higher risk myelodysplastic syndrome patients unresponsive to hypomethylating agents with ON 01910.Na. Leuk Res. 2012 Jan;36(1):98-103. doi: 10.1016/j.leukres.2011.08.022. Epub 2011 Sep 14. PMID 21924492
- [Result] Silverman LR, Greenberg P, Raza A, Olnes MJ, Holland JF, Reddy P, Maniar M, Wilhelm F. Clinical activity and safety of the dual pathway inhibitor rigosertib for higher risk myelodysplastic syndromes following DNA methyltransferase inhibitor therapy. Hematol Oncol. 2015 Jun;33(2):57-66. doi: 10.1002/hon.2137. Epub 2014 Apr 29. PMID 24777753
- [Result] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- [Derived] Navada SC, Fruchtman SM, Odchimar-Reissig R, Demakos EP, Petrone ME, Zbyszewski PS, Holland JF, Silverman LR. A phase 1/2 study of rigosertib in patients with myelodysplastic syndromes (MDS) and MDS progressed to acute myeloid leukemia. Leuk Res. 2018 Jan;64:10-16. doi: 10.1016/j.leukres.2017.11.006. Epub 2017 Nov 11. PMID 29144985